CLINICAL TRIAL: NCT02317809
Title: An Open-label, Randomized, Two-period, Two-sequence Crossover Trial to Assess the Bioequivalence of the Liquid Formulation Versus the Freeze-dried Formulation of 900 IU r-hFSH and 450 IU r-hLH in Pergoveris®, Administered Subcutaneously in Pituitary Suppressed Healthy Premenopausal Female Subjects
Brief Title: Bioequivalence Trial of Liquid Versus Freeze-Dried Pergoveris® in Pituitary Suppressed Healthy Premenopausal Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 200061-006; 2014-003506-32 (EudraCT Number)
Record Dates: First submitted 2014-12-11; First posted 2014-12-16 (Estimated); Results first posted 2016-12-13 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2017-10

CONDITIONS: Healthy
Keywords: Healthy; Pergoveris; Bioequivalence; Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- First Liquid Pergoveris, Then Freeze-dried Pergoveris (Experimental)
  Interventions: Drug: Liquid pergoveris; Drug: Freeze-dried pergoveris
- First Freeze-dried Pergoveris, Then Liquid Pergoveris (Experimental)
  Interventions: Drug: Liquid pergoveris; Drug: Freeze-dried pergoveris

INTERVENTIONS:
Drug: Liquid pergoveris — All subjects will be administered with 900 IU of r-hFSH and 450 IU of r-hLH solution (Liquid Pergoveris) as subcutaneous injection using a disposable pen-injector on Day 1 in either first intervention period or second intervention period.
Drug: Freeze-dried pergoveris — All subjects will be administered with 900 IU of r-hFSH and 450 IU of r-hLH freeze-dried powder (Freeze-dried Pergoveris) as subcutaneous injection on Day 1 in either first intervention period or second intervention period.

SUMMARY:
Some women cannot have children because they cannot produce enough follicle stimulating hormone (FSH) and luteinising hormone (LH). When this happens the ovaries fail to produce an egg during the menstrual cycle - a condition known as anovulation. Anovulation can be treated by giving replacement FSH and LH. Pergoveris is a medication that contains both FSH and LH. It is used for the treatment of anovulation in women who do not produce enough FSH and LH.

A new, liquid formulation of Pergoveris is being tested in this study. It will be compared with the current freeze-dried marketed formulation to see if the new formulation gets into the blood stream as easily as the current formulation.

This study will involve 38 healthy female subjects and 2 treatment periods and will last for approximately 77 days. Each subject will receive a single dose of the new liquid formulation and a single dose of the current marketed formulation separated by an interval of two weeks in a randomised (by chance) order. Blood samples will be taken at regular intervals over 2 weeks after each dose to measure levels of FSH and LH.

To participate female subjects must have normal ovaries on internal ultrasound scan, a normal result from a cervical smear test, be taking the combined oral contraceptive (OC) pill.

Eligible subjects will have their usual OC pill replaced with another called Marvelon throughout the study. After 14 days subjects will have their levels of FSH and LH checked and if sufficiently reduced will only then proceed to dosing.

Subjects will then receive one of the formulations. An ultrasound scan of the ovaries will be performed 7 days later, and another one 7 days later just before the next dose. Subjects whose ovaries show signs of stimulation will not be given the second dose. The ultrasound scan will be repeated 7 days after the second dose.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women aged 18 to 40 years (both inclusive) at Screening
* Taking a combined oral contraceptive (COCP) for at least 1 year prior to Screening and willing to recommence taking their own COCP from Day 43 of the Marvelon cycle until follow-up
* Normal follicle-stimulating hormone (FSH) (less than [<] 12 international units per liter [IU/L]) and estradiol levels (<100 picogram per milliliter [pg/mL])
* Gave written informed consent prior to any trial-related procedure
* Forearm veins suitable for cannulation or repeated venipuncture
* Body weight of greater than or equal to (>=) 48 kilogram (kg) and a body mass index (BMI) between 18.5 and 29.9 kilogram per square meter (kg/m^2) (both inclusive)
* Clinically acceptable values for vital signs (systolic blood pressure [SBP], diastolic blood pressure [DBP], pulse rate, and body temperature), as assessed by the Investigator
* Non-smoking or having refrained from smoking for at least 6 months prior to Screening and with a history of <10 pack years [number of pack years = (number of cigarettes per day/20)*number of years smoked]
* Able to communicate well with the Investigator, understanding the protocol requirements and restrictions, and willing to comply with the requirements of the entire trial
* Negative pregnancy test at Screening, before the start of the Marvelon cycle, and at admission (Day -1 Period 1 and Day -1 Period 2)
* Willing to use additional nonhormonal contraceptives (for example, condoms or occlusive cap [diaphragm or cervical/vault cap] with spermicide, nonhormonal intrauterine device, previous sterilization of the subject or her partner, being sexually inactive) from Day 1 of the Marvelon cycle up to follow-up
* Normal liquid-based cervical cytology assessment (Papanicolaou test score <II) within the last 12 months before Screening. If not performed as part of routine clinical care, a cervical cytology assessment must be performed as part of the Screening assessments and the result must be normal

Exclusion Criteria:

* Any surgical or medical condition, including findings in the medical history or in the pre-trial assessments, that in the opinion of the Investigator, constitutes a risk or a contraindication for the participation of the subject in the trial or that could interfere with the trial objectives, conduct, or evaluation
* Any clinically relevant abnormality in the safety laboratory parameters, as judged by the Investigator
* Any clinically significant abnormality on the 12-lead resting electrocardiogram (ECG), as judged by the Investigator
* Positive results from the serology examination for hepatitis B surface antigen, hepatitis C virus, or the human immunodeficiency virus
* Contraindications to COCP use shown by a history of conditions specified in the protocol
* History of tumors of the pituitary gland or hypothalamus
* Clinically significant abnormalities of the genital organs as determined by gynecological examination and transvaginal ultrasound (TVUS) and based on the Investigator's judgment for example, ovarian tumors, nonfunctional ovarian cysts, endometrial hyperplasia)
* Not successfully down-regulated by showing luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels above 1.0 IU/L and estradiol levels above 100 pg/mL before investigational medicinal product (IMP) administration or showing more than12 immature follicles per ovary. In that case there should be no signs of polycystic ovary syndrome (PCOS) morphology
* Polycystic ovarian syndrome as defined in the protocol
* Ovarian follicle-like structures larger than 13 millimeter (mm) during COCP use (at Screening)
* Contraindication to treatment with gonadotropins (ovarian enlargement or cyst not due to PCOS and of unknown origin, gynecological hemorrhages of unknown etiology, ovarian, uterine, or mammary carcinoma, tumors of the hypothalamus and pituitary gland, hypersensitivity to gonadotropins or to any of the excipients, extrauterine pregnancy in the previous 3 months, and medical history or risk factors for thromboembolic events)
* Pregnant or breastfeeding a child
* Prior treatment with FSH and or LH containing products
* Definite or suspected personal history or family history of an adverse drug reaction or hypersensitivity to drugs with a similar chemical structure to FSH or LH
* History or presence of asthma (with the exception of childhood asthma) or any serious allergy (requiring hospitalization or prolonged systemic treatment)
* History or presence of drug or alcohol abuse
* Positive test for drugs of abuse (including alcohol)
* Loss or donation of more than 500 mL of blood within 90 days prior to the first IMP administration
* Administration of any IMP or use of any investigational device within 60 days prior to the first IMP administration
* Use of drugs that may reduce the effectiveness of COCP from the start of the Marvelon cycle until last pharmacokinetic sample. For example, phenytoin, barbiturates, primidone, carbamazapine, oxcarbazepine, topiramate, felbamate, rifampicin, nelfinavir, ritonavir, griseofulvin, oral ketoconazole, and herbal remedies containing Hypericum perforatum (St John's Wort)
* Unlikely to comply with the protocol requirements, instructions, and trial-related restrictions for example, uncooperative attitude, inability to return for follow-up, and improbability of completing the trial
* Is (or is a relative of) the Principal Investigator or any Sub-investigator, Research Assistant, Pharmacist, Trial Coordinator, or other staff directly involved in the conduct of the trial
* Vulnerable subjects (for example, persons kept in detention)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2015-01-31 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2015-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Please contact the Merck KGaA Communication Center, Darmstadt, Germany

REFERENCES:
- [Derived] Bagchus W, Yalkinoglu O, Wolna P. Open-Label, Randomized, Two-Way, Crossover Study Assessing the Bioequivalence of the Liquid Formulation versus the Freeze-Dried Formulation of Recombinant Human FSH and Recombinant Human LH in a Fixed 2:1 Combination (Pergoveris(R)) in Pituitary-Suppressed Healthy Women. Front Endocrinol (Lausanne). 2018 Jan 11;8:371. doi: 10.3389/fendo.2017.00371. eCollection 2017. PMID 29375477

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 34 subjects were randomized and treated. Of these, 31 subjects completed the study. This was a crossover study with washout of 14 to 17 days between the two intervention periods.
Groups:
- First Liquid Pergoveris, Then Freeze-dried Pergoveris: Subjects were administered with 900 international units (IU) of recombinant human follicle-stimulating hormone (r-hFSH) and 450 IU of recombinant human luteinizing hormone (r-hLH) solution (Liquid Pergoveris) as subcutaneous injection using a disposable pen-injector on Day 1 in the first intervention period followed by 900 IU of r-hFSH and 450 IU of r-hLH freeze-dried powder (Freeze-dried Pergoveris) as subcutaneous injection on Day 1 in the second intervention period. Both the periods were separated by a washout period of 14 to 17 days.
- First Freeze-dried Pergoveris, Then Liquid Pergoveris: Subjects were administered with 900 IU of r-hFSH and 450 IU of r-hLH freeze-dried powder (Freeze-dried Pergoveris) as subcutaneous injection on Day 1 in the first intervention period followed by 900 IU of r-hFSH and 450 IU of r-hLH solution (Liquid Pergoveris) as subcutaneous injection using a disposable pen-injector on Day 1 in the second intervention period. Both the periods were separated by a washout period of 14 to 17 days.
Period: First Intervention Period (8 Days)
Arm/Group | First Liquid Pergoveris, Then Freeze-dried Pergoveris | First Freeze-dried Pergoveris, Then Liquid Pergoveris
Started | 17 | 17
Completed | 14 | 17
Not Completed | 3 | 0
Not completed — Protocol Non-Compliance | 2 | 0
Not completed — Withdrawn Due To Multiple Follicles | 1 | 0
Period: Second Intervention Period (8 Days)
Arm/Group | First Liquid Pergoveris, Then Freeze-dried Pergoveris | First Freeze-dried Pergoveris, Then Liquid Pergoveris
Started | 14 | 17
Completed | 14 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all subjects who received at least 1 dose of the investigational medicinal product (IMP) (that is, either liquid formulation or freeze-dried formulation).
Groups:
- All Subjects: All subjects who were administered with 900 IU of r-hFSH and 450 IU of r-hLH solution (Liquid Pergoveris) as subcutaneous injection using a disposable pen-injector or 900 IU of r-hFSH and 450 IU of r-hLH freeze-dried powder (Freeze-dried Pergoveris) as subcutaneous injection on Day 1 in either first or second intervention period.
Arm/Group | All Subjects
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.6 (5.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Baseline Corrected Area Under the Concentration-Time Curve From Zero to Last Quantifiable Concentration (AUC 0-t,Adj) for Follicle-Stimulating Hormone (FSH)
Description: The AUC (0-t) was defined as the area under the serum concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration. Baseline-corrected AUC0-t (AUC0-t,adj) = AUC0-t - (baseline concentration * t).
Time Frame: Pre-dose, 2, 4, 6, 7, 8, 9, 10, 12, 15, 18, 24, 36, 48, 60, 72, 96, 120 and 168 hours post-dose in each period
Population: Pharmacokinetic (PK) analysis set: All randomized subjects who were treated with both liquid and freeze-dried formulations and had absence of relevant protocol violations, had availability of the primary target variables and successfully down regulated baseline levels of FSH and LH below 1.0 IU/L in both the screening and dedicated PK assays.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: International units*hour/liter (IU*h/L)
Groups:
- Liquid Pergoveris: All subjects who were administered with 900 IU of r-hFSH and 450 IU of r-hLH solution (Liquid Pergoveris) as subcutaneous injection using a disposable pen-injector on Day 1 in either first intervention period or second intervention period.
- Freeze-dried Pergoveris: All subjects who were administered with 900 IU of r-hFSH and 450 IU of r-hLH freeze-dried powder (Freeze-dried Pergoveris) as subcutaneous injection on Day 1 in either first intervention period or second intervention period.
Arm/Group | Liquid Pergoveris | Freeze-dried Pergoveris
Number analyzed (Participants) | 22 | 22
International units*hour/liter (IU*h/L) | 3187.4 (24.3) | 2775.4 (22.0)
Statistical Analysis 1: Comparison: Liquid Pergoveris vs Freeze-dried Pergoveris; Mixed model analysis was used; Test type: Non-Inferiority or Equivalence — Bio-equivalence Analysis was performed with Equivalence Acceptance Range for 90% Confidence Interval (CI) as 80.00% - 125.00%; Geometric least squares (LS) mean ratio = 114.45, 90% CI 2-sided [110.87 to 118.15] — Percentage of geometric LS mean ratio was presented

2. Primary Outcome: Baseline Corrected Area Under the Concentration-Time Curve From Zero to Last Quantifiable Concentration (AUC0-t,Adj) for Luteinizing Hormone (LH)
Description: as for outcome 1
Time Frame: Pre-dose, 2, 4, 6, 7, 8, 9, 10, 12, 15, 18, 24, 36, 48, 60, 72, 96 and 120 hours post-dose in each period
Population: Pharmacokinetic (PK) analysis set: all randomized subjects who were treated with both liquid and freeze-dried formulations and had absence of relevant protocol violations, had availability of the primary target variables and successfully downregulated baseline levels of FSH and LH below 1.0 IU/L in both the screening and dedicated PK assays.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: International units*hour/liter (IU*h/L)
Arm/Group | Liquid Pergoveris | Freeze-dried Pergoveris
Number analyzed (Participants) | 22 | 22
International units*hour/liter (IU*h/L) | 210.4 (25.8) | 195.2 (22.5)
Statistical Analysis 1: Comparison: Liquid Pergoveris vs Freeze-dried Pergoveris; Mixed model analysis was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric least squares (LS) mean ratio = 106.99, 90% CI 2-sided [101.42 to 112.86] — Percentage of geometric LS mean ratio was presented

3. Primary Outcome: Baseline Corrected Maximum Serum Concentration (Cmax,Adj) for Follicle-Stimulating Hormone (FSH)
Description: Baseline-corrected Cmax (Cmax,adj) = Cmax - baseline concentration
Time Frame: Pre-dose, 2, 4, 6, 7, 8, 9, 10, 12, 15, 18, 24, 36, 48, 60, 72, 96, 120 and 168 hours post-dose in each period
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: International units per liter (IU/L)
Arm/Group | Liquid Pergoveris | Freeze-dried Pergoveris
Number analyzed (Participants) | 22 | 22
International units per liter (IU/L) | 47.92 (27.3) | 42.55 (29.0)
Statistical Analysis 1: Comparison: Liquid Pergoveris vs Freeze-dried Pergoveris; Mixed model analysis was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric least squares (LS) mean ratio = 112.67, 90% CI 2-sided [106.44 to 119.27] — Percentage of geometric LS mean ratio was presented

4. Primary Outcome: Baseline Corrected Maximum Serum Concentration (Cmax,Adj) for Luteinizing Hormone (LH)
Description: Baseline-corrected Cmax (Cmax,adj) = Cmax - baseline concentration.
Time Frame: Pre-dose, 2, 4, 6, 7, 8, 9, 10, 12, 15, 18, 24, 36, 48, 60, 72, 96 and 120 hours post-dose in each period
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: International units per liter (IU/L)
Arm/Group | Liquid Pergoveris | Freeze-dried Pergoveris
Number analyzed (Participants) | 22 | 22
International units per liter (IU/L) | 10.126 (31.1) | 9.782 (24.1)
Statistical Analysis 1: Comparison: Liquid Pergoveris vs Freeze-dried Pergoveris; Mixed model analysis was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric least squares (LS) mean ratio = 103.27, 90% CI 2-sided [93.16 to 114.47] — Percentage of geometric LS mean ratio was presented

5. Secondary Outcome: Baseline Corrected Area Under the Serum Concentration-time Curve From Time 0 to Infinity (AUC0-inf, Adj) for Follicle-stimulating Hormone (FSH) and Luteinizing Hormone (LH)
Time Frame: Pre-dose, 2, 4, 6, 7, 8, 9, 10, 12, 15, 18, 24, 36, 48, 60, 72, 96, 120, 168 hours post-dose in each period for FSH; Pre-dose, 2, 4, 6, 7, 8, 9, 10, 12, 15, 18, 24, 36, 48, 60, 72, 96, 120 hours post-dose in each period for LH
Population: PK analysis set. Here "n" signifies those subjects who were evaluable for the specified hormone level in each arm, respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: International units*hour/liter (IU*h/L)
Arm/Group | Liquid Pergoveris | Freeze-dried Pergoveris
Number analyzed (Participants) | 22 | 22
International units*hour/liter (IU*h/L)
  Follicle-stimulating Hormone (n=22, 22) | 3366.6 (24.2) | 2912.1 (22.2)
  Luteinizing Hormone (n=21, 22) | 216.1 (25.2) | 201.1 (21.2)

6. Secondary Outcome: Baseline Corrected Area Under the Serum Concentration-time Curve From Time Tlast Extrapolated to Infinity (%AUCextra,Adj) for Follicle-stimulating Hormone (FSH) and Luteinizing Hormone (LH)
Description: Area under the serum concentration-time curve from Tlast extrapolated to infinity given as a percentage of AUC0-inf. Data was not planned to be summarized if AUCextra,adj was less than 20%.
Time Frame: as for outcome 5
Population: As per statistical analysis plan, data was not planned to be summarized because AUCextra,adj was below 20% for all the participants.
Arm/Group | Liquid Pergoveris | Freeze-dried Pergoveris
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Apparent Terminal Elimination Rate Constant (Lambda[z]) for Follicle-stimulating Hormone (FSH) and Luteinizing Hormone (LH)
Description: The elimination rate constant was obtained from linear regression of the terminal phase of the log transformed concentration-time data.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per Hour (1/hour)
Arm/Group | Liquid Pergoveris | Freeze-dried Pergoveris
Number analyzed (Participants) | 22 | 22
Per Hour (1/hour)
  Follicle-stimulating Hormone (n=22, 22) | 0.01880 (14.2) | 0.01963 (10.0)
  Luteinizing Hormone (n=21, 22) | 0.05542 (17.1) | 0.05094 (25.5)

8. Secondary Outcome: Time to Reach the Maximum Serum Concentration (Tmax) for Follicle-stimulating Hormone (FSH) and Luteinizing Hormone (LH)
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Liquid Pergoveris | Freeze-dried Pergoveris
Number analyzed (Participants) | 22 | 22
Hour (h)
  Follicle-stimulating Hormone | 23.983 [8.23 to 36.00] | 16.575 [9.00 to 36.12]
  Luteinizing Hormone | 8.000 [6.03 to 12.00] | 7.725 [3.98 to 10.03]

9. Secondary Outcome: Apparent Terminal Half-life (t1/2) for Follicle-stimulating Hormone (FSH) and Luteinizing Hormone (LH)
Description: Terminal half-life is the time measured for the concentration to decrease by one half.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour (h)
Arm/Group | Liquid Pergoveris | Freeze-dried Pergoveris
Number analyzed (Participants) | 22 | 22
Hour (h)
  Follicle-stimulating Hormone (n=22, 22) | 36.87 (14.2) | 35.31 (10.0)
  Luteinizing Hormone (n=21, 22) | 12.507 (17.1) | 13.608 (25.5)

10. Secondary Outcome: Apparent Serum Clearance (CL/F) for Follicle-stimulating Hormone (FSH) and Luteinizing Hormone (LH)
Description: Clearance is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained is influenced by the fraction of the dose absorbed and was expressed as volume (Liter) per unit of time (hour).
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Arm/Group | Liquid Pergoveris | Freeze-dried Pergoveris
Number analyzed (Participants) | 22 | 22
Liter per hour (L/h)
  Follicle-stimulating Hormone (n=22, 22) | 0.2673 (24.2) | 0.3091 (22.2)
  Luteinizing Hormone (n=21, 22) | 2.082 (25.2) | 2.238 (21.2)

11. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz/F) for Follicle-stimulating Hormone (FSH) and Luteinizing Hormone (LH)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired concentration. Apparent volume of distribution (Vz/F) is influenced by the fraction absorbed.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Liquid Pergoveris | Freeze-dried Pergoveris
Number analyzed (Participants) | 22 | 22
Liter (L)
  Follicle-stimulating Hormone (n=22, 22) | 14.219 (27.1) | 15.742 (21.4)
  Luteinizing Hormone (n=21, 22) | 37.57 (28.8) | 43.93 (32.3)

12. Secondary Outcome: Number of Subjects With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a subject, regardless of causal relationship with the treatment. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs include both SAEs and non-serious AEs.
Time Frame: Day 1 post-IMP administration up to follow-up visit (Day 18) for IMP intervention periods
Population: as for baseline characteristics
Measure: Number; unit: Subjects
Arm/Group | Liquid Pergoveris | Freeze-dried Pergoveris
Number analyzed (Participants) | 34 | 31
Subjects
  AEs | 12 | 14
  SAEs | 1 | 0

13. Secondary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs) Related to Laboratory Assessments, Vital Signs or Electrocardiogram Findings
Time Frame: Day 1 post-IMP administration up to follow-up visit (Day 18) for IMP intervention periods
Population: as for baseline characteristics
Measure: Number; unit: Subjects
Arm/Group | Liquid Pergoveris | Freeze-dried Pergoveris
Number analyzed (Participants) | 34 | 31
Subjects | 0 | 0

14. Secondary Outcome: Number of Subjects With Follicle Size Greater Than (>)13 Millimeter
Description: Transvaginal ultrasound (TVUS) was performed to determine the follicle size and number.
Time Frame: Day 1 (pre-dose) up to follow-up visit (Day 18) for IMP intervention periods
Population: as for baseline characteristics
Measure: Number; unit: Subjects
Arm/Group | Liquid Pergoveris | Freeze-dried Pergoveris
Number analyzed (Participants) | 34 | 31
Subjects | 0 | 0

15. Secondary Outcome: Serum Estradiol Levels
Description: Data was planned to be presented as per the sequence of treatment received.
Time Frame: Screening (up to 28 days), Day 1 (pre-dose) and Day 8 in Period 1, Day 1 (pre-dose), Day 8 and follow-up (Day 18) in Period 2
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: nanogram per liter (ng/L)
Arm/Group | First Liquid Pergoveris, Then Freeze-dried Pergoveris | First Freeze-dried Pergoveris, Then Liquid Pergoveris
Number analyzed (Participants) | 17 | 17
nanogram per liter (ng/L)
  Screening (n= 17, 16) | 14.906 (9.1722) | 15.561 (4.8726)
  Period 1: Day 1 (pre-dose) (n= 16, 17) | 11.388 (3.7346) | 11.369 (2.7208)
  Period 1: Day 8 (n= 16, 17) | 11.833 (4.2363) | 12.077 (3.6155)
  Period 2: Day 1 (pre-dose) (n= 14, 16) | 12.469 (2.8548) | 11.975 (2.6377)
  Period 2: Day 8 (n= 13, 17) | 15.454 (6.6420) | 47.958 (141.2149)
  Follow-up (Day 18) (n= 16, 17) | 15.714 (7.5121) | 15.997 (6.5632)

16. Secondary Outcome: Number of Subjects With Local Tolerability/Injection Site Reactions (ISRs)
Description: Injection site was assessed by the study site staff for any local reaction (redness, swelling, bruising, and itching). Redness and bruising were scaled as None (no visible redness or bruising); Mild (less than or equal to [<=] 2.0 centimeters [cm] redness or bruising); Moderate (greater than [>] 2 to <=5.0 cm redness or bruising); Severe (>5.0 cm redness or bruising). Swelling was scaled as None (no swelling detected); Mild (palpable 'firmness' only); Moderate (<= 4 cm swelling); Severe (>4 cm swelling). Itching was scaled as None (no itching); Mild itching; Moderate itching and Severe itching. Only those scale categories which report at least 1 subject were presented.
Time Frame: 5 minutes, 1, 2, 4, 6, 12, and 24 hours post-dose in each period
Population: Safety analysis set included all subjects who received at least 1 dose of the investigational medicinal product (IMP) (that is, either liquid formulation or freeze-dried formulation). Here "n" signifies those subjects who were evaluable for the specified injection site reaction at the specified time point for each arm, respectively.
Measure: Number; unit: Subjects
Arm/Group | Liquid Pergoveris | Freeze-dried Pergoveris
Number analyzed (Participants) | 34 | 31
Subjects
  No Bruising: Day 1, 5 min (n= 34, 31) | 34 | 31
  No Bruising: Day 1, 1 hour (n= 32, 31) | 32 | 31
  No Bruising: Day 1, 2 hour (n= 34, 31) | 34 | 31
  No Bruising: Day 1, 4 hour (n= 34, 30) | 34 | 30
  No Bruising: Day 1, 6 hour (n= 33, 30) | 33 | 30
  No Bruising: Day 1, 12 hour (n= 32, 30) | 32 | 30
  No Bruising: Day 1, 24 hour (n= 34, 28) | 34 | 28
  No Itching: Day 1, 5 min (n= 34, 31) | 34 | 31
  No Itching: Day 1, 1 hour (n= 32, 31) | 32 | 31
  No Itching: Day 1, 2 hour (n= 34, 31) | 34 | 31
  No Itching: Day 1, 4 hour (n= 34, 30) | 34 | 30
  No Itching: Day 1, 6 hour (n= 33, 30) | 32 | 30
  Mild Itching: Day 1, 6 hour (n= 33, 30) | 1 | 0
  No Itching: Day 1, 12 hour (n= 32, 30) | 32 | 30
  No Itching: Day 1, 24 hour (n= 34, 28) | 34 | 28
  No Redness: Day 1, 5 min (n= 34, 31) | 30 | 26
  Mild Redness: Day 1, 5 min (n= 34, 31) | 4 | 5
  No Redness: Day 1, 1 hour (n= 32, 31) | 30 | 30
  Mild Redness: Day 1, 1 hour (n= 32, 31) | 2 | 1
  No Redness: Day 1, 2 hour (n= 34, 31) | 34 | 30
  Mild Redness: Day 1, 2 hour (n= 34, 31) | 0 | 1
  No Redness: Day 1, 4 hour (n= 34, 30) | 34 | 29
  Mild Redness: Day 1, 4 hour (n= 34, 30) | 0 | 1
  No Redness: Day 1, 6 hour (n= 33, 30) | 33 | 29
  Mild Redness: Day 1, 6 hour (n= 33, 30) | 0 | 1
  No Redness: Day 1, 12 hour (n= 32, 30) | 32 | 30
  No Redness: Day 1, 24 hour (n= 34, 28) | 34 | 28
  No Swelling: Day 1, 5 min (n= 34, 31) | 34 | 31
  No Swelling: Day 1, 1 hour (n= 32, 31) | 32 | 31
  No Swelling: Day 1, 2 hour (n= 34, 31) | 34 | 31
  No Swelling: Day 1, 4 hour (n= 34, 30) | 34 | 30
  No Swelling: Day 1, 6 hour (n= 33, 30) | 33 | 30
  No Swelling: Day 1, 12 hour (n= 32, 30) | 32 | 30
  No Swelling: Day 1, 24 hour (n= 34, 28) | 34 | 28

17. Secondary Outcome: Pain Visual Analogue Scale (VAS) Score
Description: The severity of pain was evaluated by the subject and recorded using a 100 millimeter (mm) visual analogue scale (VAS) ranging from 0 to 100, where 0 mm = no pain and 100 mm = worst possible pain.
Time Frame: 5 minutes, 1, 2, 4, 6, 12, and 24 hours post-dose in each period
Population: Safety analysis set included all subjects who received at least 1 dose of the investigational medicinal product (IMP) (that is, either liquid formulation or freeze-dried formulation). Here "n" signifies those subjects who were evaluable for the specified time point in each arm, respectively.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Liquid Pergoveris | Freeze-dried Pergoveris
Number analyzed (Participants) | 34 | 31
mm
  Day 1, 5 min (n= 34, 31) | 1.9 (4.04) | 2.5 (4.19)
  Day 1, 1 hour (n= 32, 31) | 0.2 (0.59) | 1.3 (5.01)
  Day 1, 2 hour (n= 34, 31) | 0.2 (0.52) | 0.3 (0.51)
  Day 1, 4 hour (n= 34, 30) | 0.1 (0.54) | 0.2 (0.57)
  Day 1, 6 hour (n= 33, 30) | 0.2 (0.46) | 1.0 (5.10)
  Day 1, 12 hour (n= 32, 30) | 0.2 (0.45) | 0.2 (0.48)
  Day 1, 24 hour (n= 34, 29) | 0.1 (0.24) | 0.1 (0.35)

18. Secondary Outcome: Number of Subjects With Anti-Drug Antibodies (ADAs) and Neutralizing Antibodies (NAbs) for Luteinizing Hormone (LH)
Time Frame: Day 1 pre-dose up to follow-up visit (Day 18) for IMP intervention periods
Population: as for baseline characteristics
Measure: Number; unit: Subjects
Arm/Group | Liquid Pergoveris | Freeze-dried Pergoveris
Number analyzed (Participants) | 34 | 31
Subjects
  Subjects with ADAs to LH | 0 | 0
  Subjects with Neutralizing antibodies to LH | NA — Neutralizing antibodies were not measured as there were no subjects who reported ADAs | NA — Neutralizing antibodies were not measured as there were no subjects who reported ADAs

19. Secondary Outcome: Anti-Drug Antibodies (ADAs) and Neutralizing Antibodies (NAbs) Titers for Luteinizing Hormone (LH)
Time Frame: Day 1 pre-dose up to follow-up visit (Day 18) for IMP intervention periods
Population: Data could not be collected as there were no subjects with positive results for ADAs and NAbs.
Arm/Group | Liquid Pergoveris | Freeze-dried Pergoveris
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Number of Subjects With Anti-Drug Antibodies (ADAs) and Neutralizing Antibodies (NAbs) for Follicle-stimulating Hormone (FSH)
Time Frame: Day 1 pre-dose and Day 8 post-dose for IMP intervention periods
Population: Safety analysis set included all subjects who received at least 1 dose of the investigational medicinal product (IMP) (that is, either liquid formulation or freeze-dried formulation). Here "n" signifies those subjects who were evaluable for the specified hormone level in each arm, respectively.
Measure: Number; unit: Subjects
Arm/Group | Liquid Pergoveris | Freeze-dried Pergoveris
Number analyzed (Participants) | 34 | 31
Subjects
  Day 1: Subjects with ADAs to FSH (n= 33, 31) | 2 | 1
  Day 8: Subjects with ADAs to FSH (n= 34, 31) | 2 | 1
  Day1: Subjects with NAbs to FSH (n= 34, 31) | NA — As per sponsor decision, it was decided not to evaluate the NAb due to low titers (noise) for the ADA. | NA — As per sponsor decision, it was decided not to evaluate the NAb due to low titers (noise) for the ADA.
  Day8: Subjects with NAbs to FSH (n= 34, 31) | NA — As per sponsor decision, it was decided not to evaluate the NAb due to low titers (noise) for the ADA. | NA — As per sponsor decision, it was decided not to evaluate the NAb due to low titers (noise) for the ADA.

21. Secondary Outcome: Number of Subjects With Anti-Drug Antibodies (ADAs) and Neutralizing Antibodies (NAbs) for Follicle-stimulating Hormone (FSH) at Follow-up Visit
Time Frame: At follow-up visit (Day 49)
Population: as for baseline characteristics
Measure: Number; unit: Subjects
Arm/Group | All Subjects
Number analyzed (Participants) | 34
Subjects
  Subjects with ADAs for FSH (n= 33) | 1
  Subjects with NAbs for FSH (n= 34) | NA — As per sponsor decision, it was decided not to evaluate the NAb due to low titers (noise) for the ADA.

22. Secondary Outcome: Anti-Drug Antibodies (ADAs) Titers for Follicle-stimulating Hormone (FSH)
Time Frame: Day 1 pre-dose and Day 8 post-dose for IMP intervention periods.
Population: Safety analysis set included all subjects who received at least 1 dose of the investigational medicinal product (IMP) (that is, either liquid formulation or freeze-dried formulation). Here, "Number of subjects analyzed" included those who have positive ADAs values.
Measure: Number; unit: Log Titers
Arm/Group | Liquid Pergoveris | Freeze-dried Pergoveris
Number analyzed (Participants) | 2 | 1
Log Titers
  Day 1: Subject 1 | 1.0 | 1.7
  Day 8: Subject 1 | 1.0 | 1.0
  Day 1: Subject 2 | 1.7 | NA — Only 1 subject had the positive ADAs value in Freeze-dried Pergoveris arm.
  Day 8: Subject 2 | 1.7 | NA — Only 1 subject had the positive ADAs value in Freeze-dried Pergoveris arm.

23. Secondary Outcome: Anti-Drug Antibodies (ADAs) Titers for Follicle-stimulating Hormone (FSH) at Follow-up Visit
Time Frame: At follow-up visit (Day 49)
Population: as for outcome 22
Measure: Number; unit: Log Titers
Arm/Group | All Subjects
Number analyzed (Participants) | 1
Log Titers | 1.0

24. Secondary Outcome: Neutralizing Antibodies (NAbs) Titers for Follicle-stimulating Hormone (FSH)
Time Frame: Day 1 pre-dose, Day 8 post-dose, follow-up visit (Day 49)
Population: Data could not be collected because as per spondor decision, there were no subjects evaluated for NAb due to low titers (noise) for the ADA .
Arm/Group | Liquid Pergoveris | Freeze-dried Pergoveris
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 post-IMP administration up to follow-up visit (Day 18) for IMP intervention periods
Arm/Group | Liquid Pergoveris | Freeze-dried Pergoveris
Serious Adverse Events (participants affected / at risk) | 1/34 | 0/31
Other Adverse Events (participants affected / at risk) | 12/34 | 14/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liquid Pergoveris (N=34) | Freeze-dried Pergoveris (N=31)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liquid Pergoveris (N=34) | Freeze-dried Pergoveris (N=31)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 1
Injection Site Discolouration (General disorders) | 1 | 0
Catheter Site Related Reaction (General disorders) | 1 | 4
Catheter Site Pain (General disorders) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 6 | 4
Dizziness (Nervous system disorders) | 1 | 3
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 1
Breast Tenderness (Reproductive system and breast disorders) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No